CLINICAL TRIAL: NCT03366805
Title: A Standardized Patient Education Video Program for Improvement of Post-Operative Recovery After Outpatient Upper Extremity Surgery
Brief Title: A Patient Education Video Program for Post-Operative Recovery After Upper Extremity Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Cassandra Mierisch, Orthopedic Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2266
Record Dates: First submitted 2017-11-29; First posted 2017-12-08 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Analgesics, Opioid; Orthopedic Surgery; Ambulatory Surgery; Education, Patient; Injuries and Wounds
Keywords: opioid; analgesic; ambulatory; orthopedic; surgery; patient education; video; medication diary
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: prospective, randomized clinical trial
Who Masked: Care Provider
Masking Description: Care provider is not informed of which patient education video(s) the patient was provided, unless that patient initiates a conversation with the provider regarding the video.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound Care Video (Active Comparator): Wound Care Patient Education Video
  Interventions: Behavioral: Wound Care Patient Education Video
- Pain Management Video Group (Experimental): Pain Management Patient Education Video
  Interventions: Behavioral: Pain Management Patient Education Video

INTERVENTIONS:
Behavioral: Pain Management Patient Education Video — Patient education video that were created in-house specifically for this project.
  Arms: Pain Management Video Group
Behavioral: Wound Care Patient Education Video — Patient education video that were created in-house specifically for this project.
  Arms: Wound Care Video

SUMMARY:
Adult patients undergoing elective outpatient, upper extremity, orthopedic surgeries will be randomized to view one of two educational programs: 1) a 2-video series regarding post-operative pain management or 2) a video regarding wound care and activity. The effect of this educational program on pain medications used, pain control efficacy, and other measures of satisfaction and recovery will be assessed.

DETAILED DESCRIPTION:
Four hundred (400) adult patients undergoing elective outpatient, upper extremity, orthopedic surgeries will be recruited by the surgeon-investigators. Patients will be randomized to view one of two educational programs: 1) a 2-video series regarding post-operative pain management or 2) a video regarding wound care and activity.

These patients will be encouraged to review the video online in the week before surgery. An intake enrollment form will be completed by an investigator using demographic information available in the chart.

Participants in both arms will complete their Patient Education Study Diary daily, for 7 days following their surgery. There are two versions of this diary: the Wound Education Version asks patients to report daily pain mediation use. The Pain Education Version does not include this section as patients in the pain management arm of the study record this information in their Recovery Diary.

The patient will be contacted again by phone and/or mail 1 year after surgery (12-14 months) using the contact information available in EPIC to determine the self-reported prevalence of chronic pain and pain medication use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients planning elective outpatient orthopedic surgery procedures by a Carilion Clinic hand surgeon will be eligible for the study.

Exclusion Criteria:

1. Patients unable or unwilling to provide informed consent
2. Patients unable to unwilling to participate in the trial (poor English language skills, blindness, cognitively disadvantaged, poor literacy skills, other barriers to participation)
3. Patients who are or suspect they may be pregnant.
4. Patients for whom the medical provider, in his professional judgment, does not feel that the study protocol would be appropriate. (to be tracked)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2020-06-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 15 Score | 2 days after surgery
  Score on the standardized Quality of Recovery 15 questionnaire How have you been feeling in the last 24 hours? (0 to 10, where 0= none of the time [poor] and 10=all of the time [excellent]) 0 1 2 3 4 5 6 7 8 9 10
  1. Able to breath easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with family or friends
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      Have you had any of the following in the last 24 hours? (10 to 0, where: 10=none of the time [excellent] and 0=all of the time [poor]) 10 9 8 7 6 5 4 3 2 1 0
  11. Moderate pain
  12. severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
PROMIS | 3 days after surgery
  PROMIS short forms administered on POD 3 - (GI belly pain 5a, GI nausea and vomiting 4a, Pain Intensity 3a, Pain Interference 4a, Sleep Disturbance 4a, Cognitive Function 4a)
number of narcotic pills used | 7 days after surgery
  number of narcotic pills used
daily pain level | 7 days after surgery
  0-10 rating scale
patient-reported satisfaction and feeling of control - pain management | 7 days after surgery
  Today, I feel in control of my pain management.
  1. Strongly agree
  2. Agree
  3. Neither agree nor disagree
  4. Disagree
  5. Strongly disagree
patient-reported satisfaction and feeling of control- wound care | 7 days after surgery
  Today, I feel in confident about how I am caring for my wound.
  1. Strongly agree
  2. Agree
  3. Neither agree nor disagree
  4. Disagree
  5. Strongly disagree
patient-reported satisfaction and feeling of control - pain management satisfaction | 7 days after surgery
  Today, I would rate my satisfaction with my pain control as (circle)
  1. Very satisfied
  2. Somewhat satisfied
  3. Neutral
  4. Somewhat dissatisfied
  5. Very dissatisfied
number of pain-related calls/visits to a healthcare provider | 7 days after surgery
  patient-reported
use of non-narcotic adjunct pain relief medication and modalities | 7 days after surgery
incidence of high risk activities - sedating medication polytherapy | 7 days after surgery
  combining narcotics with muscle relaxants/sedatives/alcohol, other sedating medications
incidence of high risk activities - NSAID polytherapy | 7 days after surgery
  combining prn NSAIDs with regularly dosed prescription NSAIDs
incidence of high risk activities - overdosing | 7 days after surgery
  exceeding daily recommended doses of pain medication
incidence of side effects and adverse events - Nausea/V omitting | 7 days after surgery
  Nausea/Vomiting
incidence of side effects and adverse events - Dizziness/balance problems | 7 days after surgery
  Dizziness/balance problems
incidence of side effects and adverse events - fatigue or sedation | 7 days after surgery
  fatigue or sedation
incidence of side effects and adverse events - headache | 7 days after surgery
  headache
incidence of side effects and adverse events - visual changes | 7 days after surgery
  visual changes
incidence of side effects and adverse events - stomach pain | 7 days after surgery
  stomach pain
incidence of side effects and adverse events - constipation | 7 days after surgery
  constipation
incidence of side effects and adverse events - diarrhea | 7 days after surgery
  diarrhea
incidence of side effects and adverse events - fever | 7 days after surgery
  fever
incidence of side effects and adverse events - rash | 7 days after surgery
  rash
incidence of side effects and adverse events - hives | 7 days after surgery
  hives
incidence of side effects and adverse events - swelling | 7 days after surgery
  swelling
incidence of side effects and adverse events - difficulty breathing/shortness of breath | 7 days after surgery
  difficulty breathing/shortness of breath
incidence of side effects and adverse events - heart palpitations/arrythmia/heart racing | 7 days after surgery
  heart palpitations/arrythmia/heart racing
incidence of side effects and adverse events - anaphylaxis | 7 days after surgery
  anaphylaxis
incidence of side effects and adverse events - ringing in ears | 7 days after surgery
  ringing in ears
incidence of side effects and adverse events - other | 7 days after surgery
  other
demonstrated patient knowledge | 7 days after surgery
  as measured by score on the follow-up quiz
prevalence of chronic opioid use | 1 year after surgery
  patient reported

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Mierisch, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Institute for Orthopedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT03366805/Prot_000.pdf
  • Informed Consent Form (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT03366805/ICF_001.pdf